CLINICAL TRIAL: NCT06791551
Title: Non-pharmacologial, Non-invassive Intervention Before Cardiac Surgry: a Randomized Controlled Trial
Brief Title: Non-pharmacologial, Non-invassive Intervention Before Cardiac Surgery: a Randomized Controlled Trial
Acronym: NICE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Shujuan Li, M.D., China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-2460-1
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Surgery
Keywords: cardiac surgery; cognitive function; stroke; delirium; non-invasive neuromodulation; Remote Ischemic Preconditioning
MeSH Terms: conditions — Stroke; Delirium | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active RIPC and tDCS (Active Comparator): RIPC and tDCS twice every day for 3 days before cardiac surgery
- sham RIPC and tDCS (Sham Comparator): Sham RIPC and tDCS twice every day for 3 days before cardiac surgery
  Interventions: Device: Sham (No Treatment)

INTERVENTIONS:
Device: active RIPC and tDCS — Preoperative use of a therapeutic device with sleeves fixed on the upper side of both arms, compressing the bilateral brachial arteries to 200mmHg for 5 minutes, resting for 5 minutes, repeating 5 times, recorded as 1 time, training once in the morning and afternoon each day, and continuing treatment for at least 3 days; Administer transcranial electrical stimulation, 2mA, 30min, for 3 days;
Device: Sham (No Treatment) — received sham treatment with the same appearance instrument;
  Arms: sham RIPC and tDCS

SUMMARY:
Perioperative neurological complications in cardiovascular surgical procedures are associated with a significant risk of mortality and disability. The goal of this clinical trial is to learn if ischemic preconditioning and transcranial electrical stimulation to reduce perioperative neurological complications. It will also learn about the safety of remote ischemic preconditioning and transcranial electrical stimulation before cardiac surgery. The main questions it aims to answer are "Do remote ischemic preconditioning and transcranial electrical stimulation make good effect on perioperative neurological complications?" "Are remote ischemic preconditioning and transcranial electrical stimulation safe?" Researchers will compare remote ischemic preconditioning and transcranial electrical stimulation to traditional treatment to see if remote ischemic preconditioning and transcranial electrical stimulation work to reduce perioperative neurological complications.

Participants will:Undergo remote ischemic preconditioning and transcranial electrical stimulation or sham treatment twice every day for 3 days before surgery.

Undertake psychological assessment and clinical symptom follow-up after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-80 years old;
2. Surgical patients with heart disease;
3. Elective surgery;
4. Patients identified as high-risk for postoperative neurological complications; Previous stroke history; Moderate to severe stenosis of the head and neck arteries was evaluated;
5. Be able to understand and comply with the requirements of clinical trial protocols, and voluntarily sign informed consent forms.

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of neurological complications 7 (± 3) days after cardiac surgery | From enrollment to the post-surgery within 7 (±3) days
  Lethal or non lethal stroke, coma, or motor impairment; Cognitive impairment or delirium

CONTACTS AND LOCATIONS:
Overall Officials: Shujuan Li, M.D., Study Director — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Department of Neurology, Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing,, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goede LL, Oxenford S, Kroneberg D, Meyer GM, Rajamani N, Neudorfer C, Krause P, Lofredi R, Fox MD, Kuhn AA, Horn A. Linking Invasive and Noninvasive Brain Stimulation in Parkinson's Disease: A Randomized Trial. Mov Disord. 2024 Nov;39(11):1971-1981. doi: 10.1002/mds.29940. Epub 2024 Jul 25. PMID 39051611
- [Background] Li C, Tao M, Chen D, Wei Q, Xiong X, Zhao W, Tan W, Yang J, Han Y, Zhang H, Zhang S, Liu H, Cao JL. Transcranial Direct Current Stimulation for Anxiety During Laparoscopic Colorectal Cancer Surgery: A Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e246589. doi: 10.1001/jamanetworkopen.2024.6589. PMID 38635271
- [Background] Law YM, Hsu C, Hingorani SR, Richards M, McMullan DM, Jefferies H, Himmelfarb J, Katz R. Randomized controlled trial of remote ischemic preconditioning in children having cardiac surgery. J Cardiothorac Surg. 2024 Jan 3;19(1):5. doi: 10.1186/s13019-023-02450-8. PMID 38172875
- [Background] Nyquist P, Georgakis MK. Remote ischemic preconditioning effects on brain vasculature. Neurology. 2019 Jul 2;93(1):15-16. doi: 10.1212/WNL.0000000000007724. Epub 2019 May 29. No abstract available. PMID 31142632
- [Background] Hardt JLS, Pohlmann P, Reissfelder C, Rahbari NN. Remote ischemic preconditioning for reduction of ischemia-reperfusion injury after hepatectomy: A randomized sham-controlled trial. Surgery. 2024 Feb;175(2):424-431. doi: 10.1016/j.surg.2023.09.042. Epub 2023 Nov 10. PMID 37951812